CLINICAL TRIAL: NCT02914782
Title: An Open Monocentric Observational Study to Investigate Fluid- and Electrolyte Balance in Post Cardiac-surgery Patients in the ICU
Brief Title: Investigation of Fluid- and Electrolyte Balance in Post Cardiac-surgery Patients
Acronym: Clinibil
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: B. Braun Melsungen AG (Industry); Center for Biomarker Research in Medicine (Unknown)
Responsible Party: Sponsor
Other Study IDs: 4947261
Record Dates: First submitted 2016-09-19; First posted 2016-09-26 (Estimated); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Electrolyte Imbalances; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Biospecimen Retention: Samples Without DNA — In the course of the stay at the ICU we will collect serum and urine samples during routine patient care to analyze for electrolytes, oxygen and kidney biomarkers.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Observational Study

SUMMARY:
Critically ill patients need intravenous fluid therapy in order to correct or prevent problems with their fluid and/or electrolyte status and for renal protection. The decision for the optimal composition and amount of IV-fluids can be difficult and complex. It is well known that errors in fluid- and electrolyte management contribute to overall morbidity and mortality. For decades, urinary sodium was used to diagnose renal disease. Nevertheless, renal excretion of sodium is largely impaired in critically ill patients, particularly in patients with acute kidney injury. Due to the high frequent measurement of renal output, it would be possible to measure the urinary electrolytes and its relative changes. Urinary electrolyte measurement may alert for the presence of the development of an akute kidney injury before occurring increases in creatinine or oliguria. The rationale of this investigation is therefore to collect data related to fluid- and electrolyte management from critically ill patients in order to find patterns of fluid- and electrolyte imbalances which may lead to disturbances and further, may allow an early detection of acute kidney injury.

DETAILED DESCRIPTION:
Critically ill patients need intravenous fluid therapy in order to correct or prevent problems with their fluid and/or electrolyte status and for renal protection. The decision for the optimal composition and amount of IV-fluids can be difficult and complex. It is well known that errors in fluid- and electrolyte management contribute to overall morbidity and mortality.

Due to the administration of large volumes of normal saline and/or a decreased urinary output of sodium or chloride iatrogen electrolyte disorders, such as hyperchloremic acidosis or dysnatremia are common abnormalities in the clinical practice. The common fact that normal saline has non-physiological levels of chloride and sodium, intensifies this problem with high volume administration. (Burdett et al. 2003; Adrogué & Madias 1997).

Hypernatremia is an independent risk factor for mortality in critically ill patients and increases the length of ICU stay (Lindner et al. 2010; Stieglmair et al. 2013) Hypernatremia is associated with impaired renal fluid regulation, as well as a lack of thirst mechanisms. In the ICU this fact requires exact measurement of all fluid- and electrolyte intake and (non-)renal losses. (Lindner et al. 2009). Therefore, in critical care settings measuring fluid balance (the difference between infusion input and renal / non-renal losses) is daily routine. The renal output is measured frequently by the nursing staff. An automated acquisition of the urinary output combined with the data of the infusion site would reduce the workload of the staff and would allow visualization of the fluid status.

Furthermore, beyond volume, the concentration and composition of the fluid is an important parameter. The comparison of urinary electrolytes with the electrolyte input from infusions allows an early detection of electrolyte disorders (Besen et al. 2015). Sodium and chloride are the main ions of solutions infused into critically ill patients. The excessive infusion of fluids lead to sodium and chloride overloads and is associated with higher mortality (Noritomi et al. 2009). For decades, urinary sodium was used to diagnose renal disease. Nevertheless, renal excretion of sodium is largely impaired in critically ill patients, particularly in patients with acute kidney injury. Due to the high frequent measurement of renal output, it would be possible also to measure the urinary electrolytes and its relative changes which are likely to be more relevant than the absolute electrolyte concentrations. Urinary electrolyte measurement may alert for the presence of AKI development before occurring increases in creatinine or oliguria (Maciel 2013; Maciel et al. 2015; Molitoris 2013).

The rationale of this investigation is therefore to collect data related to fluid- and electrolyte management from critically ill patients in order to find patterns of fluid- and electrolyte imbalances which may lead to disturbances and further, may allow an early detection of acute kidney injury (AKI).

Patients undergoing scheduled cardiac surgery will be included in this trial. The rationale behind this is on the one hand, that the patient cohort is homogenous and on the other hand, that the risk for developing an AKI is 30-40% among cardiac surgery patients (Rosner et al. 2006). The aim is to detect characteristic patterns in electrolyte metabolism between patients who develop an AKI and those who do not.

ELIGIBILITY:
Inclusion Criteria:

i. 8 years or older ii. Expected length of stay at the ICU > 48 hours iii. eGFR (CKD-EPI) > 45 ml/min iv. ACR < 300 mg/g creatinine v. signed informed consent prior to cardiac surgery

Exclusion Criteria:

i. renal insufficiency (eGFR-CKD-EPI < 45 ml/min), dialysis ii. severe infection (fever > 38 °C, CRP > 50 ml/l) iii. increased risk for perioperative multi-organ failure due to co-morbidities such as cardiogenic decompensation pre-surgery, low cardiac output, incipient cardiogenic shock and sepsis iv. Karnofsky Index < 40 v. hearing impairment vi. physical and mental illnesses vii. missing signed informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 adult patients (<18 years, m&f) will be included in this study. All patients will be assigned with randomized numbers to stay anonymous. Patients scheduled for cardiac-surgery with normal renal function will be included to assure a homogenous clinical picture. These patients will be transferred to the intensive care unit post-surgery where electrolyte and fluid data will be collected along with serum and urine samples. The will remain in the study only during their stay at the ICU.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2022-10 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
Routine laboratory measurements and ELISA to define urinary and serum biomarkers for the early diagnosis of acute kidney injury. | 1 year
  Serum and urine will be collected multiple times daily and analyzed for Na, K, Osmolality, Cl and oxygen concentration. Serum and urine ELISA assays will be carried out to detect changes in concentration of KIM-1, NGAL, Cystatin-C and E-Selectin.

SECONDARY OUTCOMES:
Measurement of fluid input and output (ml) to define trends in electrolyte and fluid balance using electronic data from ICU | 1 year
  Define how renal status correlates with the electrolyte balance of the patient by analyzing trend curves of fluid input (ml of infusion solution, ml parenteral nutrition, etc.) and output (ml urine, ml drainages, etc.) over the course of the stay at the ICU. The data will be entered manually into a software program routinely used at the ICU.

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Eller, MD Prof, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

REFERENCES:
- [Background] Besen BA, Gobatto AL, Melro LM, Maciel AT, Park M. Fluid and electrolyte overload in critically ill patients: An overview. World J Crit Care Med. 2015 May 4;4(2):116-29. doi: 10.5492/wjccm.v4.i2.116. eCollection 2015 May 4. PMID 25938027
- [Background] Stieglmair S, Lindner G, Lassnigg A, Mouhieddine M, Hiesmayr M, Schwarz C. Body salt and water balances in cardiothoracic surgery patients with intensive care unit-acquired hyponatremia. J Crit Care. 2013 Dec;28(6):1114.e1-5. doi: 10.1016/j.jcrc.2013.05.017. Epub 2013 Jul 24. PMID 23890940
- [Background] Lindner G, Kneidinger N, Holzinger U, Druml W, Schwarz C. Tonicity balance in patients with hypernatremia acquired in the intensive care unit. Am J Kidney Dis. 2009 Oct;54(4):674-9. doi: 10.1053/j.ajkd.2009.04.015. Epub 2009 Jun 10. PMID 19515476
- [Background] Maciel AT. Breaking old and new paradigms regarding urinary sodium in acute kidney injury diagnosis and management. Crit Care. 2013 Feb 4;17(1):115. doi: 10.1186/cc11926. PMID 23384365
- [Background] Molitoris BA. Measuring glomerular filtration rate in the intensive care unit: no substitutes please. Crit Care. 2013 Sep 4;17(5):181. doi: 10.1186/cc12876. PMID 24004539
- [Background] Maciel AT, Nassar AP Jr, Vitorio D. Very Transient Cases of Acute Kidney Injury in the Early Postoperative Period After Cardiac Surgery: The Relevance of More Frequent Serum Creatinine Assessment and Concomitant Urinary Biochemistry Evaluation. J Cardiothorac Vasc Anesth. 2016 Jan;30(1):56-63. doi: 10.1053/j.jvca.2015.04.020. Epub 2015 Apr 28. PMID 26296826
- [Background] Adrogue HJ, Madias NE. Aiding fluid prescription for the dysnatremias. Intensive Care Med. 1997 Mar;23(3):309-16. doi: 10.1007/s001340050333. PMID 9083234
- [Background] Noritomi DT, Soriano FG, Kellum JA, Cappi SB, Biselli PJ, Liborio AB, Park M. Metabolic acidosis in patients with severe sepsis and septic shock: a longitudinal quantitative study. Crit Care Med. 2009 Oct;37(10):2733-9. doi: 10.1097/ccm.0b013e3181a59165. PMID 19885998
- [Background] Rosner MH, Okusa MD. Acute kidney injury associated with cardiac surgery. Clin J Am Soc Nephrol. 2006 Jan;1(1):19-32. doi: 10.2215/CJN.00240605. Epub 2005 Oct 19. PMID 17699187